CLINICAL TRIAL: NCT02991768
Title: Budesonide for Mycophenolic Acid (MPA)-Induced Diarrhea in Renal Transplant Recipients
Brief Title: Budesonide for Mycophenolic Acid-induced Diarrhea in Renal Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment not continued
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00140436
Record Dates: First submitted 2016-11-21; First posted 2016-12-13 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Entocort EC (Experimental): Subjects will take 6mg Entocort EC by mouth daily for 8 weeks.
  Interventions: Drug: Entocort
- Placebo (Placebo Comparator): Subjects will take 6mg matching placebo pill daily for 8 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Entocort — A corticosteroid that decreases levels of inflammatory cytokines.
  Other Names: budesonide
  Arms: Entocort EC
Drug: Placebos — Placebo is matched to the study drug.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn if using a Entocort (budesonide) to treat diarrhea will be effective and safe for kidney transplant patients, allowing them to continue with MPA medication.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients > 1 months post-transplant,
* No history of chronic diarrhea pre-transplant,
* >3 watery/soft stools after transplant on at least 4 days in the week without anti-diarrheal for at least 2 weeks or using anti-diarrheals for at least 4 days in the week > 2 weeks
* Subjects on at least 180mg twice a day of mycophenolate-sodium or 250 mg twice a day of cellcept

Exclusion Criteria:

* Diagnosis of any known colonic diseases (i.e. Crohn's disease, ulcerative colitis, ischemic colitis, Celiac disease), partial colonic resection, small bowel resection, history of cholecystectomy, Irritable Bowel Syndrome, fecal Incontinence, Bacterial overgrowth, infectious diarrhea (c difficle, cryptospora, giardia, isospora, Human Immunodeficiency Virus), Cytomegalovirus colitis
* Subjects with recent acute rejection treated with high dose steroids
* Subjects taking Boswellia serrata extract, over-the-counter herbs, cholestyramine, nonsteroidal salicylates (other than daily ASA)
* Subjects with active malignancy, liver cirrhosis, active peptic ulcer disease, known intolerance or resistance to budesonide, pregnancy, breast-feeding, mental retardation
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Budhiraja, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Entocort EC
Started | 9
Completed | 5
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Entocort EC
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 48.3 [26 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission of Diarrhea
Description: Measured using symptom diary. Complete remission (CR) is defined as a mean of <3 stools/day and a mean of <1 watery stool per day without use of anti-diarrheal drugs.
Time Frame: Week 8
Population: Data not collected. Physician left the institution and study was terminated.
Arm/Group | Entocort EC
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS)
Description: GSRS is a 15-item instrument designed to assess the symptoms associated with common GI disorders. The GSRS consists of 5 subscales (reflux, diarrhea, constipation, abdominal pain, and indigestion) producing a mean subscale score ranging from 1 (no discomfort) to 7 (very severe discomfort).
Time Frame: Change from Baseline to Week 8
Population: Data not collected. Physician left the institution and study was terminated.
Arm/Group | Entocort EC
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS)
Description: as for outcome 2
Time Frame: Change from Baseline to Week 16
Population: Data not collected. Physician left the institution and study was terminated.
Arm/Group | Entocort EC
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Gastrointestinal Quality of Life Index (GIQLI)
Description: The GIQLI is a 36-item questionnaire to assess the impact of GI disease on daily life. The GIQLI has 5 subscales (GI symptoms, emotional status, physical functions, social functions, and stress of medical treatment), producing a total score of the 36 items. Lower scores represent more dysfunction.
Time Frame: Change from Baseline to Week 8
Population: Data not collected. Physician left the institution and study was terminated.
Arm/Group | Entocort EC
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Gastrointestinal Quality of Life Index (GIQLI)
Description: as for outcome 4
Time Frame: Change from Baseline to Week 16
Population: Data not collected. Physician left the institution and study was terminated.
Arm/Group | Entocort EC
Number analyzed (Participants) | 0

6. Secondary Outcome: MPA Dose
Time Frame: Change from Baseline to Week 8
Population: Data not collected. Physician left the institution and study was terminated.
Arm/Group | Entocort EC
Number analyzed (Participants) | 0

7. Secondary Outcome: MPA Dose
Time Frame: Change from Baseline to Week 16
Population: Data not collected. Physician left the institution and study was terminated.
Arm/Group | Entocort EC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of study participation - 16 weeks.
Arm/Group | Entocort EC
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT02991768/Prot_SAP_001.pdf